CLINICAL TRIAL: NCT02490826
Title: Intervention Software for Children With Speech Sound Disorders
Brief Title: Table to Tablet (T2T): A Novel Intervention Framework for Children With Speech Sound Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Luís Miguel Teixeira de Jesus, Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PGIS73
Record Dates: First submitted 2015-06-22; First posted 2015-07-07 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Speech Disorders
Keywords: Speech Sound Disorders; Tabletop; Digital
MeSH Terms: conditions — Speech Disorders; Speech Sound Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Table-based T2T intervention (Active Comparator): A combined phonological awareness therapy, listening and discrimination and auditory bombardment activities intervention will be applied. This will be based in a table top material version.
  The intervention will consist of 12 weekly sessions (individual) of 45 min in duration, divided into two blocks (6+6) without any breaks.
  Interventions: Other: Table-based T2T intervention
- Tablet-based T2T intervention (Active Comparator): A combined phonological awareness therapy, listening and discrimination and auditory bombardment activities intervention will be applied. This will be based in a tablet (digital) material version.
  The intervention will consist of 12 weekly sessions (individual) of 45 min in duration, divided into two blocks (6+6) without any breaks.
  Interventions: Other: Tablet-based T2T intervention

INTERVENTIONS:
Other: Table-based T2T intervention — Phonological therapy consists of a combination of phonological awareness activities, auditory and discrimination and auditory bombardment activities. This activities will be based on table top materials. The items used in the intervention will be based on the child's target speech production goals. This intervention will include the following areas:
  * Auditory Bombardment;
  * Auditory and discrimination;
  * Letter-sound knowledge;
  * Phoneme identity and phoneme matching;
  * Blending;
  * Segmentation;
  * Rhyme;
  * Phoneme manipulation.
  Arms: Table-based T2T intervention
Other: Tablet-based T2T intervention — Phonological therapy consists of a combination of phonological awareness activities, auditory and discrimination and auditory bombardment activities. This activities will be based on digital materials presented on a tablet. The items used in the intervention will be based on the child's target speech production goals. This intervention will include the following areas:
  * Auditory Bombardment;
  * Auditory and discrimination;
  * Letter-sound knowledge;
  * Phoneme identity and phoneme matching;
  * Blending;
  * Segmentation;
  * Rhyme;
  * Phoneme manipulation.
  Arms: Tablet-based T2T intervention

SUMMARY:
The primary aim of this study is to develop software as a tool in speech and language therapy for the treatment of children (Portuguese and English) with phonologically based Speech Sound Disorders (SSD). Further, this project aims to test the effectiveness of this approach with two groups of preschool and school aged children with phonologically based SSD, with one group consisting of European Portuguese (EP) speakers and one group of British English (BE) speakers. Performance across the two groups will be compared. The total duration of the project will be 30 month.

DETAILED DESCRIPTION:
The Table to Tablet (T2T) project aims to develop software as a tool in speech and language therapy for the treatment of children (Portuguese and English) with phonologically based Speech Sound Disorders (SSD). Further, this project aims to test the effectiveness of this approach with two groups of children aged between 3 years and 6 months and 6 years and 6 months with phonologically based Speech Sound Disorders (SSD).

One group consists of European Portuguese (EP) speakers and one group of British English (BE) speakers. Each group should include 20 children with the referred criteria and the performance across the two groups will be compared.

The total duration of the project will be 30 month (software development over the first 12 months and an intervention study during following 18 months).

The T2T team includes 3 Speech and Language Therapists and 3 engineers/researchers plus a designer that will develop the T2T material.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of Phonologically based Speech and Sound Disorder;
* Portuguese as native language;
* Audition of 20 decibels (dB) or lower in the frequencies 500, 1000, 2000 and 4000;
* Normal non-verbal ability (NVIQ) according to age;
* Receptive language skills within normal limits.

Exclusion Criteria:

* Diagnose of childhood apraxia of speech;
* Structural or functional oral alterations

Ages: 42 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-10; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Consonants Correct | one year
  Calculation of the percentage of the correct produced consonants

SECONDARY OUTCOMES:
Parental Reports | one and a half year
  Questionnaire focused on: speech improvement; enjoyment of therapy; effect of therapy on their understanding of their child.
Intelligibility Score | one year
  How well a client's speech is understood by other individuals, i.e. understandability of speech.
Percentage of occurence of phonological processes | one year
  Calculations of the percentage of occurence of phonological processes
Generalisation Score | one year
  Generalization probe of the trained phonological process to five non-intervention words.
Phonetic Inventory | one year
  List of produces consonants
Percentage of Correct Vowels | one year
  Calculation of the percentage of the correct produced vowels
Percentage of Phonemes Correct | one year
  Calculation of the percentage of the correct produced phonemes

CONTACTS AND LOCATIONS:
Overall Officials: Luís MT Jesus, Principal Investigator — Aveiro's University
Locations (1):
- Aveiro's University, Aveiro, Portugal

REFERENCES:
- [Background] Lousada M, Jesus LM, Capelas S, Margaca C, Simoes D, Valente A, Hall A, Joffe VL. Phonological and articulation treatment approaches in Portuguese children with speech and language impairments: a randomized controlled intervention study. Int J Lang Commun Disord. 2013 Mar-Apr;48(2):172-87. doi: 10.1111/j.1460-6984.2012.00191.x. Epub 2012 Dec 4. PMID 23472957
- [Background] Lousada M, Jesus LM, Hall A, Joffe V. Intelligibility as a clinical outcome measure following intervention with children with phonologically based speech-sound disorders. Int J Lang Commun Disord. 2014 Sep-Oct;49(5):584-601. doi: 10.1111/1460-6984.12095. Epub 2014 May 26. PMID 24861159
- [Derived] Jesus LM, Santos J, Martinez J. The Table to Tablet (T2T) Speech and Language Therapy Software Development Roadmap. JMIR Res Protoc. 2019 Jan 30;8(1):e11596. doi: 10.2196/11596. PMID 30698534
- See also: Official T2T website — http://t2t.web.ua.pt/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT02490826/Prot_SAP_000.pdf